CLINICAL TRIAL: NCT07204509
Title: Incidence of Chromosomal Abnormalities in Patients With Congenital Heart Diseases Attending Assiut University Children's Hospital
Brief Title: Chromosomal Abnormalities in Patients With Congenital Heart Disease at Assiut University Children's Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alyaa Ramadan Ibrahim, Resident, pediatrics Department, Assiut University
Other Study IDs: AUN-CHD-Genetics-2025
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Congenital Heart Disease (CHD); Chromosomal Abnormalities
Keywords: Karyotyping; gentic disease
MeSH Terms: conditions — Heart Defects, Congenital; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Congenital Heart Disease: This cohort includes pediatric patients with a confirmed diagnosis of congenital heart disease (CHD) attending Assiut University Children's Hospital and Elmabara Insurance Hospital. All participants underwent clinical evaluation, dysmorphic feature assessment, and cytogenetic testing (karyotyping) to detect chromosomal abnormalities. No therapeutic interventions were applied as part of this study; data were collected for observational and genetic analysis purposes only.
  Interventions: Diagnostic Test: Conventional Karyotyping

INTERVENTIONS:
Diagnostic Test: Conventional Karyotyping — Conventional chromosomal analysis was performed using karyotyping of peripheral blood lymphocytes. Standard cytogenetic techniques were applied to identify chromosomal abnormalities in pediatric patients with congenital heart disease. This diagnostic test was used solely for observational and genetic correlation purposes.

SUMMARY:
Congenital heart disease (CHD) is one of the most common birth defects and an important cause of infant morbidity and mortality. Many children with CHD also have underlying genetic abnormalities, particularly chromosomal abnormalities, which may affect their prognosis, management, and counseling. This study aims to determine the incidence and pattern of chromosomal abnormalities among children with CHD attending Assiut University Children's Hospital and Elmabara Insurance Hospital.

Children with a confirmed diagnosis of CHD will undergo a detailed clinical assessment, including dysmorphic evaluation, followed by chromosomal analysis (karyotyping). The study will help identify the frequency and type of chromosomal abnormalities associated with CHD and their correlation with specific cardiac defects and phenotypic features.

Understanding these genetic associations may improve diagnosis, early intervention, and family counseling, and provide useful information for risk stratification and prevention strategies in the Egyptian population.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) affects approximately 8-10 per 1,000 live births worldwide. Genetic factors, including chromosomal abnormalities such as trisomies and microdeletions, are strongly associated with the occurrence of CHD. Identifying such abnormalities is important for patient management, surgical planning, long-term prognosis, and genetic counseling.

This observational cross-sectional study will be conducted at Assiut University Children's Hospital (Pediatric Genetics Unit and Pediatric Cardiology Clinic) and Elmabara Insurance Hospital. A total of 138 children with confirmed structural CHD will be enrolled. Each patient will undergo:

Clinical evaluation including demographic data, detailed medical history, and physical examination.

Assessment of dysmorphic features and other congenital anomalies.

Cytogenetic evaluation using standard karyotyping to detect chromosomal abnormalities.

The primary outcome is to estimate the incidence of chromosomal abnormalities in children with CHD. Secondary outcomes include the correlation of specific chromosomal abnormalities with CHD subtypes and phenotypic features.

This study will contribute valuable data regarding the genetic background of CHD in Upper Egypt. The findings are expected to enhance the understanding of genotype-phenotype correlations, improve early diagnosis, and guide family counseling and preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Children with a confirmed diagnosis of congenital heart disease (by echocardiography and/or cardiology evaluation).
* Age between 1 month and 18 years.
* Patients attending Assiut University Children's Hospital or Elmabara Insurance Hospital during the study period.
* Informed consent obtained from parents or legal guardians.

Exclusion Criteria:

* Patients with acquired (non-congenital) heart disease.
* Critically ill patients in unstable condition not suitable for blood sampling.
* Incomplete clinical data or refusal of parents/guardians to participate.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study population consists of pediatric patients with congenital heart disease attending Assiut University Children's Hospital and Elmabara Insurance Hospital. Eligible children underwent detailed clinical evaluation, dysmorphic assessment, and cytogenetic testing (karyotyping) to determine the incidence and pattern of chromosomal abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Chromosomal Abnormalities among Children with Congenital Heart Disease | At enrollment (karyotype performed at baseline during the study period: September 2025 - September 2026)
  Proportion of enrolled pediatric CHD patients with any chromosomal abnormality detected by conventional karyotyping of peripheral blood lymphocytes. Chromosomal abnormalities include numerical (e.g., trisomies, monosomies) and large structural rearrangements visible on karyotype.
Incidence of Chromosomal Abnormalities among Children with Congenital Heart disease | At enrollment (karyotype performed at baseline during the study period: october 2025 - October 2026)
  Proportion of enrolled pediatric CHD patients with any chromosomal abnormality detected by conventional karyotyping of peripheral blood lymphocytes. Chromosomal abnormalities include numerical (e.g., trisomies, monosomies) and large structural rearrangements visible on karyotype.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] S. Zaidi and M. Brueckner, "CHD Epidemiology: Evidence for Genetics Underlying CHD Congenital Heart Disease Compendium Genetics and Genomics of Congenital Heart Disease," 2017,
- [Background] Wang H, Lin X, Lyu G, He S, Dong B, Yang Y. Chromosomal abnormalities in fetuses with congenital heart disease: a meta-analysis. Arch Gynecol Obstet. 2023 Sep;308(3):797-811. doi: 10.1007/s00404-023-06910-3. Epub 2023 Jan 7. PMID 36609702
- [Background] Pierpont ME, Brueckner M, Chung WK, Garg V, Lacro RV, McGuire AL, Mital S, Priest JR, Pu WT, Roberts A, Ware SM, Gelb BD, Russell MW; American Heart Association Council on Cardiovascular Disease in the Young; Council on Cardiovascular and Stroke Nursing; and Council on Genomic and Precision Medicine. Genetic Basis for Congenital Heart Disease: Revisited: A Scientific Statement From the American Heart Association. Circulation. 2018 Nov 20;138(21):e653-e711. doi: 10.1161/CIR.0000000000000606. PMID 30571578